CLINICAL TRIAL: NCT01173380
Title: Effects of Soy on Metabolite Markers of Health
Brief Title: Soy Nut Study on Markers of Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200715715-4
Record Dates: First submitted 2010-07-23; First posted 2010-08-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome X
Keywords: Soy; Equol; Metabolic syndrome; Endothelial function
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matched food (Sham Comparator): Control food (matched for calories and macronutrients) per day for 4 weeks
  Interventions: Other: Matched food
- Soy nuts (Active Comparator): Oil roasted soy nuts with 101 milligrams of soy isoflavones per day for 4 weeks
  Interventions: Other: Soy nuts

INTERVENTIONS:
Other: Soy nuts — Oil roasted soy nuts with 101 milligrams of soy isoflavones per day for 4 weeks
  Other Names: Genisoy
  Arms: Soy nuts
Other: Matched food — Control food (matched for calories and macronutrients) per day for 4 weeks
  Arms: Matched food

SUMMARY:
The investigators hope to learn about the effects of soy nuts on markers of health. When some people eat soy foods, their gut bacteria make equol. Equol is a soy metabolite (small molecule made during metabolism). The investigators will be testing blood samples to determine if markers of health are different for people who make equol versus people who do not make equol.

DETAILED DESCRIPTION:
The objective of the study is to investigate the metabolomic response to consumption of soy protein containing polyphenolic phytochemicals (isoflavones). The aim of this pilot study is to demonstrate proof of concept and ability to detect metabolomic changes that are responsive to soy. This preliminary data will then be used to design future research projects.

Food phytochemicals such as the polyphenolic flavonoids from a wide variety of foods and beverages have been associated with cardiovascular protective effects in epidemiologic studies. Significant controversy exists in the literature regarding the efficacy and mechanisms for the cardiovascular protection of soy foods. The soy hypothesis for cardiovascular risk reduction has been focused mainly on the isoflavone content of soy, but uncertainty still exists regarding the bioactive component(s). In particular, consumption of soy protein foods has been associated with favorable cardiovascular disease (CVD) risk profiles in population based studies. Controlled clinical trials and meta-analyses however, have resulted in the conclusions that soy protein with associated isoflavones has only modest hypocholesterolemic effects in the range of 3-5% reduction in LDL-cholesterol. Additional cardioprotective effects have been demonstrated in clinical trials, promoting small but significant changes in vascular endothelial function and antioxidant protection. An important observation is that animal studies have shown reduction in atherosclerotic lesion size both with and without decreased blood lipid levels. These results taken together suggest that soy and soy phytochemicals can promote positive risk factors and outcomes by mechanisms in addition to, and other than lowering serum cholesterol levels. There is a need for greater understanding of the cellular and molecular mechanisms underlying the physiologic responses to isoflavones in the vascular compartment. Increasing evidence is emerging that biologically relevant concentrations of isoflavones may impact cell signaling processes in vascular and other tissues.

The large body of literature on human clinical trials of soy proteins and isoflavones has focused primarily on traditional lipid and lipoprotein parameters, biomarkers of CVD risk, and functional changes in endothelial function, platelet activation and total blood antioxidant capacity as described above. It is possible and likely that the effect of soy consumption on CVD risk is a net result of multiple subtle changes in metabolic pathways, vascular inflammatory responses and cell-signaling pathways which are not readily detected in healthy individuals. Since individuals with metabolic syndrome (MetS) present with many of the metabolic aberrations purported to be improved through soy food ingestion, these individuals may be an excellent study population in order to investigate the effects of a soy food intervention on metabolic markers of health. Equol is the end-product of daidzein biotransformation, and is produced only by some humans, resulting in a phenotypic characteristic in response to dietary soy. It is hypothesized by some researchers that the "equol producers" may have additional metabolic and phenotypic responses to soy which may help to explain some of the variances in the literature. Few investigators have examined this question in existing studies, with two reporting an association with outcomes and one no association. A recent study using microarray analysis of lymphocytes from postmenopausal women demonstrated differential gene expression in women who form equol compared to those who do not, suggesting that equol status may be an important modulator of responses to soy isoflavones. No studies have examined this question in a metabolomic investigation. This demonstrates a gap in the literature and provides an opportunity to contribute significant novel data using cutting-edge approaches.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Men ages 45 or above
* Blood pressure greater than or equal to 130/85 mmHg but not greater than 160/100 and meeting an additional 2 of the remaining 4 Metabolic syndrome diagnostic criteria as defined by NCEP ATP III:

  1. Elevated waist circumference: men equal to or greater than 40 inches, women equal to or greater than 35 inches
  2. Reduced HDL cholesterol: men less than 40 mg/dL, women less than 50 mg/dL
  3. Fasting glucose greater than or equal to 100 mg/dL
  4. Fasting blood triglycerides greater than or equal to 150 mg/dL but less than 400 mg/dL
* Weight of at least 110 pounds

Exclusion Criteria:

* Smokers
* Chronic disease, such as diabetes, cancer, renal disease, and blood disorders
* History of intestinal disorders, which affect absorption or transit, such as ulcerative colitis or crohns disease
* Allergy to soy
* Antioxidant supplement usage

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Improve lipid profile | After 4 week intervention
  Total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglyceride level, apolipoproteinA1, apolipoproteinB100, apolipoproteinB100:apolipoproteinA1, urinary F2-isoprostane
Increase endothelial function | After 4 week intervention
  Brachial artery flow mediated dilation, reactive hyperemia peripheral arterial tonometry, blood pressure, endothelin-1
Attenuate glycemic responses | After 4 week intervention
  Fasting plasma glucose, insulin, fructosamine, homeostasis model assessment of insulin resistance

SECONDARY OUTCOMES:
Decrease inflammatory markers | After 4 week intervention
  High sensitivity C reactive protein, vascular cell adhesion molecule-1, intercellular adhesion molecule-1
Follow anthropometrics for stable weight | After 4 week intervention
  Weight, height, body mass index, waist circumference, hip circumference, waist:hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Francene M Steinberg, PhD, RD, Principal Investigator — UC Davis
Locations (1):
- Ragle Human Nutrition Center, Davis, California, United States

REFERENCES:
- [Background] Azadbakht L, Kimiagar M, Mehrabi Y, Esmaillzadeh A, Hu FB, Willett WC. Soy consumption, markers of inflammation, and endothelial function: a cross-over study in postmenopausal women with the metabolic syndrome. Diabetes Care. 2007 Apr;30(4):967-73. doi: 10.2337/dc06-2126. PMID 17392557
- [Background] Azadbakht L, Kimiagar M, Mehrabi Y, Esmaillzadeh A, Padyab M, Hu FB, Willett WC. Soy inclusion in the diet improves features of the metabolic syndrome: a randomized crossover study in postmenopausal women. Am J Clin Nutr. 2007 Mar;85(3):735-41. doi: 10.1093/ajcn/85.3.735. PMID 17344494
- [Background] Bartoli G, Menegaz G, Lisi M, Di Stolfo G, Dragoni S, Gori T. Model-based analysis of flow-mediated dilation and intima-media thickness. Int J Biomed Imaging. 2008;2008:738545. doi: 10.1155/2008/738545. Epub 2009 Apr 6. PMID 19360110
- [Background] Bitto A, Altavilla D, Bonaiuto A, Polito F, Minutoli L, Di Stefano V, Giuliani D, Guarini S, Arcoraci V, Squadrito F. Effects of aglycone genistein in a rat experimental model of postmenopausal metabolic syndrome. J Endocrinol. 2009 Mar;200(3):367-76. doi: 10.1677/JOE-08-0206. Epub 2008 Dec 9. PMID 19066292
- [Background] Cassidy A, Brown JE, Hawdon A, Faughnan MS, King LJ, Millward J, Zimmer-Nechemias L, Wolfe B, Setchell KD. Factors affecting the bioavailability of soy isoflavones in humans after ingestion of physiologically relevant levels from different soy foods. J Nutr. 2006 Jan;136(1):45-51. doi: 10.1093/jn/136.1.45. PMID 16365057
- [Background] Charles C, Yuskavage J, Carlson O, John M, Tagalicud AS, Maggio M, Muller DC, Egan J, Basaria S. Effects of high-dose isoflavones on metabolic and inflammatory markers in healthy postmenopausal women. Menopause. 2009 Mar-Apr;16(2):395-400. doi: 10.1097/gme.0b013e3181857979. PMID 18981951
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] de Kleijn MJ, van der Schouw YT, Wilson PW, Grobbee DE, Jacques PF. Dietary intake of phytoestrogens is associated with a favorable metabolic cardiovascular risk profile in postmenopausal U.S.women: the Framingham study. J Nutr. 2002 Feb;132(2):276-82. doi: 10.1093/jn/132.2.276. PMID 11823590
- [Background] Donald AE, Halcox JP, Charakida M, Storry C, Wallace SM, Cole TJ, Friberg P, Deanfield JE. Methodological approaches to optimize reproducibility and power in clinical studies of flow-mediated dilation. J Am Coll Cardiol. 2008 May 20;51(20):1959-64. doi: 10.1016/j.jacc.2008.02.044. PMID 18482664
- [Background] Grundy SM. Metabolic syndrome pandemic. Arterioscler Thromb Vasc Biol. 2008 Apr;28(4):629-36. doi: 10.1161/ATVBAHA.107.151092. Epub 2008 Jan 3. PMID 18174459
- [Background] Hallund J, Bugel S, Tholstrup T, Ferrari M, Talbot D, Hall WL, Reimann M, Williams CM, Wiinberg N. Soya isoflavone-enriched cereal bars affect markers of endothelial function in postmenopausal women. Br J Nutr. 2006 Jun;95(6):1120-6. doi: 10.1079/bjn20061734. PMID 16768834
- [Background] Kreijkamp-Kaspers S, Kok L, Bots ML, Grobbee DE, Lampe JW, van der Schouw YT. Randomized controlled trial of the effects of soy protein containing isoflavones on vascular function in postmenopausal women. Am J Clin Nutr. 2005 Jan;81(1):189-95. doi: 10.1093/ajcn/81.1.189. PMID 15640479
- [Background] Kressel G, Trunz B, Bub A, Hulsmann O, Wolters M, Lichtinghagen R, Stichtenoth DO, Hahn A. Systemic and vascular markers of inflammation in relation to metabolic syndrome and insulin resistance in adults with elevated atherosclerosis risk. Atherosclerosis. 2009 Jan;202(1):263-71. doi: 10.1016/j.atherosclerosis.2008.04.012. Epub 2008 Apr 20. PMID 18501910
- [Background] Li SH, Liu XX, Bai YY, Wang XJ, Sun K, Chen JZ, Hui RT. Effect of oral isoflavone supplementation on vascular endothelial function in postmenopausal women: a meta-analysis of randomized placebo-controlled trials. Am J Clin Nutr. 2010 Feb;91(2):480-6. doi: 10.3945/ajcn.2009.28203. Epub 2009 Nov 18. PMID 19923372
- [Background] Maskarinec G, Steude JS, Franke AA, Cooney RV. Inflammatory markers in a 2-year soy intervention among premenopausal women. J Inflamm (Lond). 2009 Apr 7;6:9. doi: 10.1186/1476-9255-6-9. PMID 19348684
- [Background] Kelm M. Flow-mediated dilatation in human circulation: diagnostic and therapeutic aspects. Am J Physiol Heart Circ Physiol. 2002 Jan;282(1):H1-5. doi: 10.1152/ajpheart.2002.282.1.H1. No abstract available. PMID 11748041
- [Background] Nasca MM, Zhou JR, Welty FK. Effect of soy nuts on adhesion molecules and markers of inflammation in hypertensive and normotensive postmenopausal women. Am J Cardiol. 2008 Jul 1;102(1):84-6. doi: 10.1016/j.amjcard.2008.02.100. Epub 2008 Apr 16. PMID 18572041
- [Background] Pipe EA, Gobert CP, Capes SE, Darlington GA, Lampe JW, Duncan AM. Soy protein reduces serum LDL cholesterol and the LDL cholesterol:HDL cholesterol and apolipoprotein B:apolipoprotein A-I ratios in adults with type 2 diabetes. J Nutr. 2009 Sep;139(9):1700-6. doi: 10.3945/jn.109.109595. Epub 2009 Jul 15. PMID 19605528
- [Background] Potenza MV, Mechanick JI. The metabolic syndrome: definition, global impact, and pathophysiology. Nutr Clin Pract. 2009 Oct-Nov;24(5):560-77. doi: 10.1177/0884533609342436. PMID 19841245
- [Background] Setchell KD, Brown NM, Lydeking-Olsen E. The clinical importance of the metabolite equol-a clue to the effectiveness of soy and its isoflavones. J Nutr. 2002 Dec;132(12):3577-84. doi: 10.1093/jn/132.12.3577. PMID 12468591
- [Background] Thorp AA, Howe PR, Mori TA, Coates AM, Buckley JD, Hodgson J, Mansour J, Meyer BJ. Soy food consumption does not lower LDL cholesterol in either equol or nonequol producers. Am J Clin Nutr. 2008 Aug;88(2):298-304. doi: 10.1093/ajcn/88.2.298. PMID 18689364
- [Background] Rufer CE, Maul R, Donauer E, Fabian EJ, Kulling SE. In vitro and in vivo metabolism of the soy isoflavone glycitein. Mol Nutr Food Res. 2007 Jul;51(7):813-23. doi: 10.1002/mnfr.200700013. PMID 17579888
- [Background] Torres N, Torre-Villalvazo I, Tovar AR. Regulation of lipid metabolism by soy protein and its implication in diseases mediated by lipid disorders. J Nutr Biochem. 2006 Jun;17(6):365-73. doi: 10.1016/j.jnutbio.2005.11.005. Epub 2005 Dec 5. PMID 16481155
- [Background] van Ee JH. Soy constituents: modes of action in low-density lipoprotein management. Nutr Rev. 2009 Apr;67(4):222-34. doi: 10.1111/j.1753-4887.2009.00192.x. PMID 19335716
- [Background] Welty FK, Lee KS, Lew NS, Zhou JR. Effect of soy nuts on blood pressure and lipid levels in hypertensive, prehypertensive, and normotensive postmenopausal women. Arch Intern Med. 2007 May 28;167(10):1060-7. doi: 10.1001/archinte.167.10.1060. PMID 17533209